CLINICAL TRIAL: NCT01227863
Title: Randomized Clinical Trial Of Drug Topics Efficacy Maxinom® (Dexamethasone + Neomycin Sulfate + Polymyxin B Sulfate - Lab. Union Chemical) And Maxitrol® (Dexamethasone + Neomycin Sulfate + Polymyxin B Sulfate - Lab. Alcon) In Reducing The Signs And Symptoms Of Acute Bacterial Conjunctivitis
Brief Title: Efficacy Maxinom® And Maxitrol® in Reducing The Signs And Symptoms Of Acute Bacterial Conjunctivitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clínica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DNPUNI0610; Version 01
Record Dates: First submitted 2010-10-15; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Bacterial Conjunctivitis; Acute
Keywords: SIGNS AND SYMPTOMS OF ACUTE BACTERIAL CONJUNCTIVITIS
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Maxitrol

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Test (Experimental): Dexamethasone + neomycyn + polimixyn B
  Interventions: Drug: MAXINOM®
- Comparator (Active Comparator): Dexamethasone + neomycyn + polimixy B
  Interventions: Drug: Maxitrol®

INTERVENTIONS:
Drug: MAXINOM® — Dexamethasone...............................................0,1% Neomicyn......................................0,35% polimixyn B...................................0,1%
  Arms: Test
Drug: Maxitrol® — Dexamethasone...............................................0,1% Neomicyn......................................0,35% Polimixyn B...................................0,1%
  Arms: Comparator

SUMMARY:
The primary objective of this study is to evaluate, through clinical parameters, the effectiveness of your medicine topic Maxinom ® (dexamethasone, neomycin and polymyxin B - Union Chemicals), comparing it to the topical medication Maxitrol ® (dexamethasone, neomycin and polymyxin B - Alcon ) by the percentage of improvement (sustained response rate) at the end of treatment, among the products studied.

DETAILED DESCRIPTION:
1. Evaluation of isolated signs and symptoms during treatment, with a record of individual scores for each parameter and observation
2. Statistical comparison of drug safety, by recording qualitative and quantitative parameters related to adverse effects occurring during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree with all study procedures and sign, by his own free will, IC;

  * Adult patients, regardless of gender, ethnicity or social status, with good mental health;
  * Patients who present at screening visit, picture of acute bacterial conjunctivitis diagnosed clinically.

Exclusion Criteria:

* Patients with clinical diagnosis or suspicion of conjunctivitis due to any process that is not due to bacterial infection, such as infections by fungi, protozoa, viruses and allergic conjunctivitis;

  * Patients with known hypersensitivity to any component of the formulas of the study drugs;
  * Patients with a history or clinical diagnosis of other lesions that may affect the outcome, such as glaucoma, corneal ulcer or scars;
  * Concomitant use of ocular medication other than the study;
  * Pregnant or lactating women;
  * Being or having been treated for any type of conjunctivitis within 15 days and have finished treatment or less than 07 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Compared effectiveness between drugs using percentage of improvement (sustained response rate) at the end of treatment. | 7 dyas of treatment.
  There will be a total of three returns after inclusion (0 day), and they are 1, 3 and 7 days after initiation of treatment. At the returns of 1 and 3 days there will be a tolerance of + 1 day and the return of 7 day, the tolerance will be +- 1 day. On each return will be collected data on the efficacy and safety.

SECONDARY OUTCOMES:
Evaluation of signs and symptoms during treatment with a record of individual scores for each parameter established. | 7 days of treatment.
  There will be a total of three returns after inclusion (0 day), and they are 1, 3 and 7 days after initiation of treatment. At the returns of 1 and 3 days there will be a tolerance of + 1 day and the return of 7 day, the tolerance will be +- 1 day. On each return will be collected data on the efficacy and safety.
Statical comparison of drug safety by recording qualitative and quantitative parameter related to adverse effects occurring during treatment. | 7 days of treatment.
  There will be a total of three returns after inclusion (0 day), and they are 1, 3 and 7 days after initiation of treatment. At the returns of 1 and 3 days there will be a tolerance of + 1 day and the return of 7 day, the tolerance will be +- 1 day. On each return will be collected data on the efficacy and safety.

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil